CLINICAL TRIAL: NCT05734768
Title: Impact of Preterm Birth on Symptoms of Anxiety and Depression in Parents, and on the Precursors of Cognition, Including Social Cognition in Their Child
Acronym: PréDANPa
Status: Recruiting | Type: Observational
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PA23021*
Record Dates: First submitted 2023-02-09; First posted 2023-02-21 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Parental Anxiety Following Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preterm newborns and their parents: Thirty premature children born between 32 and 36+6 weeks of gestation, and their parents.
  Interventions: Behavioral: State-Trait Anxiety Inventory - Y ou STAI-Y
- term newborns and their parents: Thirty children, born at more than 37 weeks (≥37+0), and their parents
  Interventions: Behavioral: State-Trait Anxiety Inventory - Y ou STAI-Y

INTERVENTIONS:
Behavioral: State-Trait Anxiety Inventory - Y ou STAI-Y — Questionnaire

SUMMARY:
In 2018, the World Health Organization (WHO) counted no less than 15 million preterm births each year worldwide, or more than one in ten children. In recent years, the number of newborns surviving preterm birth has gradually increased due to advances in neonatal medicine. However, these rescues are not without consequences.

Indeed, to do so, the child is separated from his parents, placed in a stressful, technical and potentially painful environment. This early separation is compounded by medical co-morbidities and sedations that compromise the child's physiology and availability to interact. Extreme prematurity also disrupts the early interactions between the child and his parents, and eventually the relationships with others. Thus, more than 35% of children born prematurely show insecure attachment behavior in their relationships with others.

Moreover, premature births are accompanied by numerous somatic, cognitive and social cognitive difficulties. At school age, these children present more learning, social-emotional and behavioral problems. The greater the degree of prematurity, the more marked these difficulties are. They would be associated with an executive and social cognition deficit, inherent to a globally altered cerebral development, in particular the frontal subcortical cerebral regions.

On the parents' side, premature birth is also fraught with consequences. Indeed, the idea of an idealized post-natal period gives way to an anxious, even traumatic experience. Notions of guilt are often expressed, as well as major anxiety about the child's survival and "parenting skills". A higher prevalence of signs of parental anxiety, postnatal depression and post-traumatic stress disorder is observed in mothers of premature infants, even up to 18 months after birth. These psychological states influence the parents' ability to interact with their newborn, as well as the content of these interactions.

Finally, both parents and newborns see, for different reasons, their ability to interact and to reassure themselves profoundly disrupted by premature birth.

Even if since 2010, prematurity has been identified as a "public health problem" by the WHO, studies on the subject still have limitations. Indeed, if we estimate that the prevalence of anxiety and/or depression signs in mothers of premature babies is on average three times higher than in mothers of full-term babies; what about fathers? It seems fundamental to improve our knowledge of the anxious and depressive symptoms that fathers and mothers of premature babies may display, with the aim of providing comprehensive and multidisciplinary care for families in neonatal intensive care units.

Similarly, the exact impact of an increase in parental anxious depressive symptomatology on the precursors of cognitive and social cognitive development is not known. Since the environment and stimulation are fundamental to the child's development, what happens when one or both parents have their interaction modified by anxious-depressive symptomatology? Indeed, the rare studies publishing data on the subject are carried out on populations of parents of non-premature children, often non-French-speaking and above all with tools that are not available to French-speaking practitioners in charge of the early detection of developmental difficulties in premature children. Today, it seems necessary to provide data concerning the development of precursors to cognitive and social cognitive development in preterm infants, and to better understand the extent of its interaction with the anxious depressive symptomatology of the mother and father.

The investigators therefore formulate the following hypotheses:

* Anxious depressive symptomatology, such as signs of parental anxiety, postnatal depression, and posttraumatic stress disorder, would be higher in mothers and fathers of preterm infants than in mothers and fathers of full-term infants at 7 ± 1 weeks after birth.
* The level of development of the precursors to cognitive and social cognitive development would be lower in children whose parents present an exacerbated anxious depressive symptomatology.

ELIGIBILITY:
Inclusion Criteria:

Children and their parents will be included in the study in the exposed group if:

* the infant is born preterm, i.e., between 32 weeks of amenorrhea (SA) and 36 SA + 6 days.
* at the maternity ward of the University Hospital of Reims
* the parents are older than 18 years.
* parents are affiliated to a social insurance.
* parents agreed to participate in the study, within 72 hours after birth

Will be included in the study, in the non-exposed group, children and their parents, if:

* the children is born at term, i.e., from 37 SA + 0 Days
* at the maternity ward of the Reims University Hospital
* parents are older than 18 years.
* parents are affiliated to a social insurance.
* parents agreed to participate in the study, within 72 hours after birth

Exclusion Criteria:

Will not be included in the study, children and their parents, if:

* the infant is born from multiple pregnancy
* the infant is hemodynamically unstable
* the birth occured more than 72 hours ago
* the infant is affected by congenital malformations
* the infant is affected by severe brain lesion detected by transfontanellar ultrasound scan performed before inclusion (cystic leukomalacia, and stages III and IV of the Papille classification i.e. severe ventricular dilatation or intra-parenchymal hemorrhage)
* separation from the parents and placement of the child is intended
* child is born anounymously
* parents with psychiatric disorders
* if the mother is suffering from hemodynamic compromise
* parents under guardianship
* parents non-native speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants included will be children born preterm (32 - 37 SA) and their parents, and children born at term and their parents, who meet the inclusion criteria and who have accepted to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-11-28 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2028-05-28 (Estimated)

PRIMARY OUTCOMES:
STAI-Y : State Trait Inventory Anxiety - Y | week 7 weeks post partum
  used to compare level of anxiety and depression in mothers of infants born preterm (32 to 37 gestational age) vs mothers of infants born at term (37 to 41 gestational age)

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France